CLINICAL TRIAL: NCT06100757
Title: Ventricular Mechanical Impact, Contraction Efficiency and Heart Function With Right Ventricular Pacing by MICRATMTPS. Comparison With Conventional RV Pacing
Brief Title: Effect of Leadless Pacing on Heart Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S59717
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Pacing-Induced Cardiomyopathy
Keywords: leadless pacemaker; Micra Transcatheter pacemaker; ventricular function; valve function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional pacing (Active Comparator): 24 patients underwent the implantation of a conventional VVI pacing system (Medtronic) with placement of a ventricular pacing lead Medtronic 5076-58 in the right ventricle.
  Interventions: Device: Conventional pacemaker type Medtronic Advisa ADSR03 or Azure XT VR
- leadless pacing (Experimental): 27 patients underwent the implantation of a leadless pacing system Micra TPS
  Interventions: Device: Micra Transcatheter Pacing System (TPS°

INTERVENTIONS:
Device: Micra Transcatheter Pacing System (TPS° — Implantation of a leadless pacemaker type Micra TPS. Echocardiographic and clinical follow-up during 12 months
  Arms: leadless pacing
Device: Conventional pacemaker type Medtronic Advisa ADSR03 or Azure XT VR — Implantation of a conventional ventricular pacemaker (VVI and VV(R) pacing mode) and right ventricular lead (Medtronic 5076-58)/ Echocardiographic and clinical follow-up during 12 months
  Arms: Conventional pacing

SUMMARY:
This prospective, un-blinded, randomized, noninferiority, single centre study with 12 month follow-up included patients who were scheduled for a single-chamber PM implant. Patients were 1:1 randomized to undergo the implantation of a conventional VVI pacing system (Medtronic, Advisa ADSR03) with a ventricular pacing lead (Medtronic, 5076-58) in the right ventricle (called 'conventional group') or to be implanted with a leadless Micra TPS (called 'Micra group').

The primary objective was to assess and compare the mechanical impact of right ventricular pacing using the Micra TPS versus a conventional PM on the left ventricular function.

DETAILED DESCRIPTION:
The primary endpoint was to assess the mechanical impact of the Micra TPS on the left ventricular function. The investigators measured the change of Global Longitudinal Strain (GLS) over one year after pacemaker implantation.

As secondary endpoint, the investigators studied the effect of the Micra TPS on the right ventricle using speckle tracking for 2-D myocardial motion estimation. The investigators also assessed conventionally the function of the right ventricle using tricuspid annular plane systolic excursion (TAPSE) in accordance with the guidelines of the European Association of Cardiovascular Imaging and American Society of Echocardiography. Evolution of clinical and biological parameters as NYHA (New York Heart Association) classification, '6 minutes 'walk distance and measurement of brain natriuretic peptide (NT-proBNP) test was also be performed at baseline and after one year follow-up.

Design

It was an interventional prospective not blinded randomized single centre study. The investigators randomized fifty patients into two groups (1:1 ratio) between May 2018 and December 2021:

Group 1 : 25 patients underwent the implantation of a conventional ventricular pacemaker (Medtronic) with placement of a ventricular lead Medtronic 5076-58 in the right ventricle.

Group 2 : 25 patients underwent the implantation of a leadless pacing system Micra TPS.

All implantation procedures were performed under local anaesthesia. To minimize the impact of the pacing site, the investigators targeted as first position the mid septum of the right ventricle. In the presence of inacceptable electrical measurements, an apical positioning was reached. All pacing positions were reviewed according to the Lieberman criteria.

Patients follow-up Patients were followed for a minimal period of 1 year (at 1 month after implantation, 6 months and 12 months as in routine care). Two-dimensional echocardiography was performed 1 day before implantation and at each visit. A 6 minutes' walk distance was performed at day 10 and at 1 year follow-up. As biological marker of the left ventricular function, brain natriuretic peptide (NT-proBNP) was also measured at baseline and at 1 year follow-up.

Device data collections:

The implant procedure duration as the procedure fluoroscopy times were also recorded. Follow-up of the electrical measurements was performed at the same time than the echocardiographic recording.

All complications (implantation failure, device or lead dislodgements, implantation related infection, death) were also prospectively documented.

Conventional 2D-Echocardiography:

Transthoracic echocardiography was performed using a commercially available ultrasound machine (VividTM E95, GE Vingmed Ultrasound AS; Epiq, Philips Medical Systems). Baseline and follow-up echocardiographic examinations were performed using the same machine. Conventional echocardiographic data were analysed according to the recommendations of the European Association of Cardiovascular Imaging. Standard parasternal long- and short-axis and apical four and two-chamber and long axis view were acquired. Left ventricular end-diastolic volume (LVEDV), end-systolic volume (LVESV) and left ventricular ejection fraction were calculated using Simpson's rule in a four-chamber view.

The ystolic function of the right ventricle was evaluated by tricuspid annular plane systolic excursion (TAPSE) in a standard apical four-chamber view. Finally, valve function and particularly tricuspid function was assessed following the European recommendations.

All echocardiographic values will be obtained from the average of measurements from six continuous normal cardiac beats.

Ethical considerations:

The investigators followed the declaration of Helsinki regarding human experimentation. Moreover, the investigators respected national legislation regarding clinical research and confidentiality of the data obtained in this study. All the participants were informed about the aims and procedures of the study and signed an informed consent form before the inclusion in the study. The local ethical committees reviewed and approved this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a Class I or II indication for single chamber pacemaker following international guidelines

Exclusion Criteria:

* patients with previously implanted cardiac devices / mechanical valves that would interfere with the echocardiographic measurements
* patients with inadequate image quality at baseline that prohibited the assessment of myocardial mechanics using echocardiography
* patients with a left ventricular ejection fraction (LVEF) ≤40% at baseline
* patients considered to have a pre-existing condition challenging/precluding the implant of a conventional pacemaker
* patients who refused or were not able to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment and comparison of the mechanical impact of right ventricular pacing using the Micra TPS versus a conventional PM on the left ventricular function. | 1 year
  The primary endpoints were the change in left ventricular ejection fraction (LVEF) and global longitudinal strain (GLS)

SECONDARY OUTCOMES:
Evolution of the right ventricular, tricuspid valve and mitral valve function | 1 year
  Echocardiographic measurements at baseline and 1-year follow-up
Evolution of NT-pro-BNP | 1 year
  Measurement of NT-pro BNP at baseline and 1-year follow-up
Evolution of pacemaker performance | 1 year
  Measurement of electrical parameters: pacing threshold, impedance and R-wave sensing. Measurement of percentage of ventricular pacing in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Garweg, MD, PhD, Principal Investigator — University hospitals of Leuven
Locations (1):
- University Hospitals of Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garweg C, Duchenne J, Vandenberk B, Mao Y, Ector J, Haemers P, Poels P, Voigt JU, Willems R. Evolution of ventricular and valve function in patients with right ventricular pacing - A randomized controlled trial comparing leadless and conventional pacing. Pacing Clin Electrophysiol. 2023 Dec;46(12):1455-1464. doi: 10.1111/pace.14870. Epub 2023 Nov 13. PMID 37957879